CLINICAL TRIAL: NCT03469037
Title: Effects on an Experimental Dyspnea by Thoraco-abdominal Elastic Strapping of the High Flow Nasal Cannula
Brief Title: Effects on Experimental Dyspnea of High Flow Nasal Cannula
Acronym: EDEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association pour le Développement et l'Organisation de la Recherche en Pneumologie et sur le Sommeil (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-A00178- 47
Record Dates: First submitted 2018-02-25; First posted 2018-03-19 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Dyspnea; Healthy Volunteers
Keywords: Dyspnea, High flow nasal cannula
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxygen first (Experimental): Optiflow with an inspired fraction of oxygen of 100% in the first seance Optiflow with an inspired fraction of oxygen of 21 % in the second seance
  Interventions: Device: Optiflow with an inspired fraction of oxygen of 100%; Device: Optiflow with an inspired fraction of oxygen of 21%
- Air first (Experimental): Optiflow with an inspired fraction of oxygen of 21 % in the first seance Optiflow with an inspired fraction of oxygen of 100 % in the second seance
  Interventions: Device: Optiflow with an inspired fraction of oxygen of 100%; Device: Optiflow with an inspired fraction of oxygen of 21%

INTERVENTIONS:
Device: Optiflow with an inspired fraction of oxygen of 100% — Respiratory gaz heated and humidified system of delivery with a fraction of oxygen inspired of 100%
  Other Names: High flow nasal cannula with oxygen added
Device: Optiflow with an inspired fraction of oxygen of 21% — Respiratory gaz heated and humidified system of delivery with a fraction of oxygen inspired of 21%
  Other Names: High flow nasal cannula without oxygen added

SUMMARY:
To develop an experimental model of dyspnea by external thoraco-abdominal elastic strapping at rest in order to study the mechanisms involved in the relief of dyspnea by the administration of high flow by nasal cannula (HFNC).

DETAILED DESCRIPTION:
This study will measure the effect of HFNC on an experimental model of dyspnea induced by thoraco-abdominal elastic strapping on healthy subjects at rest.

The study will also compare the effects on dyspnea of the administration of high flow nasal cannula with and without oxygen added.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* chronic pathology
* active smokers
* anxiety disorder
* allergy to latex
* protected adult
* woman declared herself pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2018-11-02 (Actual)

PRIMARY OUTCOMES:
Effects of high flow nasal cannula on strapping induced type of dyspnea | One hour
  Evaluated by visual annylogic scale

SECONDARY OUTCOMES:
Compare the effect of the high flow by nasal cannula with and without oxygen on an experimental dyspnea, evaluated by the differences of changes in the visual analogic scale | One hour
  Evaluated by visual annylogic scale

CONTACTS AND LOCATIONS:
Overall Officials: Capucine Morelot-Panzini, Doctor, Principal Investigator — Service de Pneumologie de la Pitié-Salpétrière; Thomas Similowski, PHD, Study Director — Service de Pneumologie de la Pitié-Salpétrière
Locations (2):
- France (2):
  - Laboratoire de Physiopathologie Respiratoire du Service de Pneumologie et de Réanimation, Paris
  - Service de Pneumologie et Réanimation Médicale, Paris

IPD SHARING:
Plan to Share IPD: No